CLINICAL TRIAL: NCT06220825
Title: PRactice of VENTilation in Critically Ill PEDiatric Patients (PRoVENT-PED) - an International Multicenter Observational Study
Brief Title: PRactice of VENTilation in Critically Ill PEDiatric Patients
Acronym: PRoVent-PED
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Other Study IDs: PRoVent-PED
Record Dates: First submitted 2024-01-08; First posted 2024-01-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Critical Illness; Respiratory Failure
Keywords: Ventilation practice; Critically ill children; PARDS; Mechanical ventilation
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this worldwide observational study is to investigate ventilation practice in critically ill pediatric patients. The main questions it aims to answer are:

1. What is the global current practice of ventilatory support in critically ill pediatric patients?
2. Which potentially modifiable factors related to ventilation are associated with outcome? Participating pediatric intensive care units will gather detailed information about ventilation practice and outcome, such as duration of ventilatory support, length of ICU stay and ICU mortality.

DETAILED DESCRIPTION:
Rationale:

Studies on ventilatory support in critically ill pediatric patients remain scarce and much of the current clinical practice is based upon experience and data originating from critically ill adult patients.

Objectives:

1. To describe the worldwide practice of ventilatory support in critically ill pediatric patients; and
2. To identify potentially modifiable ventilation parameters that have independent associations with outcome.

Hypothesis:

1. Practice of ventilatory support in critically ill pediatric patients varies substantially worldwide; and
2. Potentially modifiable factors related to ventilation have independent associations with outcome in critically ill pediatric patients.

Study design:

International, multicenter, observational cohort study in critically ill pediatric patients. Each year, data will be collected in two predefined 4-week periods, one in the winter season and one in the summer season. A third 4-week period will be in case of epi- or pandemics. The study is designed to run for 10 years; within these 10 years, there will be subprojects during pre-defined periods. Centers have the option to opt out during certain time periods to make the study manageable for every participating country/center.

Study population:

Critically ill pediatric patients (aged 0-18) admitted to the pediatric intensive care unit (PICU) and necessitating ventilatory support > 12 hours. Premature infants will be excluded. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Because of the observational design of the study using routinely collected data, there is no additional burden for the patient. Collection of data from ICU charts or electronic medical records systems is of no risk to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Expected use of (non-)invasive respiratory support for at least 12 hrs

Exclusion Criteria:

* premature infants (i.e., postconceptional age corrected for gestational age < 40 weeks)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Critically ill pediatric patients
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2034-04-01 (Estimated); Study Completion 2034-04-01 (Estimated)

PRIMARY OUTCOMES:
Tidal volume | First four days of (non-)invasive respiratory support
  Tidal volume
Peak inspiratory pressure | First four days of (non-)invasive respiratory support
  Peak inspiratory pressure
Plateau pressure | First four days of (non-)invasive respiratory support
  Pateau pressure
Positive end-expiratory pressure | First four days of (non-)invasive respiratory support
  Positive end-expiratory pressure
Driving pressure | First four days of (non-)invasive respiratory support
  Driving pressure
Mechanical power | First four days of (non-)invasive respiratory support
  Mechanical power

SECONDARY OUTCOMES:
PARDS prevalence | First four days of (non-)invasive respiratory support
  Prevalence of PARDS per PALICC-2 definition
Duration of respiratory support (in days) | Up to 28 days following initiation of (non-)invasive respiratory support
  Duration of respiratory support (in days)
Ventilator-free days at day 28 | Up to 28 days following initiation of (non-)invasive respiratory support
  Ventilator-free days at day 28
Length of ICU stay (in days) | PICU admission
  Length of ICU stay (in days)
ICU mortality | Up to 28 days following initiation of (non-)invasive respiratory support
  ICU mortality

OTHER OUTCOMES:
Type of ventilatory support | First four days of (non-)invasive respiratory support
  Type of ventilatory support
Type of ventilator mode | First four days of (non-)invasive respiratory support
  Ventilator mode
Use of sedative and/or analgesic drugs (yes/no) | First four days of (non-)invasive respiratory support
  Use of sedative and/or analgesic drugs
Use of neuromuscular blocking agents (yes/no) | First four days of (non-)invasive respiratory support
  Use of neuromuscular blocking agents
Use of vasoactive infusions (yes/no) | First four days of (non-)invasive respiratory support
  Use of vasoactive infusions
Use of prone positioning (yes/no) | First four days of (non-)invasive respiratory support
  Use of prone positioning
Use of ECMO (yes/no) | First four days of (non-)invasive respiratory support
  Use of ECMO

CONTACTS AND LOCATIONS:
Overall Officials: Martin CJ Kneyber, MD PhD, Principal Investigator — University Medical Center Groningen; Marcus J Schultz, MD PhD, Principal Investigator — Amsterdam UMC; Frederique Paulus, RN PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- UMC Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: PRoVent-PED study website — https://icuresearch.nl/studies/provent-ped